## Exploring the optimal timing of minimally invasive surgery for esophageal squamous cell carcinoma after neoadjuvant chemoradiotherapy

October 15, 2021

## **Statistical Analysis**

The Fisher's exact test was used to compare categorical data. Survival analysis was performed using the Kaplan–Meier method. Multivariable analyses using logistic regression and Cox proportional hazards models were performed to derive odds ratios (OR) and hazard ratios (HR) as effect-size measures, with 95% CIs. Statistical significance was set at p<0.05 for all analyses.

Data analysis was conducted using R version 3.5.3 (R Foundation for Statistical Computing, Vienna, Autria). The full R code to train the models is available supplementary, along with a list of packages used.